CLINICAL TRIAL: NCT05473975
Title: Search for a Recanalization of the Sylvian Artery Electro-Physiological Biomarker
Acronym: BEERS
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MOA_2022_3
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: AIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Placement of the EGG — Placement of the EGG before the beginning of the thrombectomy

SUMMARY:
Early recanalization is a major prognostic factor in vascular accidents ischemic brain injury (AIC). The acute phase therapies of AIC aim to recanalization by intravenous thrombolysis and/or mechanical thrombectomy. Recanalization is identified immediately during thrombectomy by per-procedural arteriography. For the thrombolysis, only a performed MRI will validate the recanalization. This "proof of concept" study aims to identify an Electro-Encephalographic biomarker (EEG) of the recanalization in real time, the EEG being easy to set up. This biomarker will be sought during recanalization certified by thrombectomy in order to identify the window time for which the biomarker must be sought on the EEG. During this study, the identified EEG biomarker can be used to validate the recanalization during the intravenous thrombolysis in future studies

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Presenting a cerebral infarction with proximal occlusion of the sylvian artery requiring thrombectomy
* No objection to participation in the study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient benefiting from legal protection
* Absence of affiliation to a social protection scheme
* Recent cranial surgery not allowing the installation of a scalp EEG

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inclusions 15 patients hospitalized for an ischemic stroke for whom an MRI identified a proximal sylvian artery occlusion, treatable by mechanical thrombectomy.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
IElectro-Encephalographic (EEG) marker of recanalization | inclusion visit
  dentification of an Electro-Encephalographic (EEG) marker of recanalization in patients with cerebral infarction with proximal occlusion of the sylvian artery and recanalized by mechanical thrombectomy

CONTACTS AND LOCATIONS:
Overall Officials: Michael OBADIA, Principal Investigator — HOPITAL FONDATION Adolphe de ROTHSCHILD
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No